CLINICAL TRIAL: NCT02171598
Title: Randomised, Open Label, 3-way Cross Over Phase I Study to Investigate the Impact of Concomitant Use of Multiple Doses of Clopidogrel (75 mg qd After a Loading Dose of 300 mg) With Multiple Doses of Dabigatran Etexilate (150 mg Bid) on the Pharmacokinetic and Pharmacodynamic Parameters, and Additionally the Impact of Single Oral Doses of 300 mg and 600 mg of Clopidogrel Administered Under Steady State Conditions of Dabigatran of 75 mg and 150 mg in Healthy Male Subjects
Brief Title: Investigation of the Impact of Concomitant Use of Multiple Doses of Clopidogrel With Multiple Doses of Dabigatran Etexilate on the Pharmacokinetic and Pharmacodynamic Parameters in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.83
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel; Dabigatran

ARMS (3):
- Fixed sequence 1 (Experimental): multiple-dose, fixed-sequence with 2 periods of 4 days separated by a washout period of at least 14 days. A single dose of 300 mg clopidogrel will be given on top of 75 mg or 150 mg dabigatran in steady state.
  Interventions: Drug: Clopidogrel; Drug: Dabigatran high dose; Drug: Dabigatran low dose
- Crossover (Experimental): clopidogrel + dabigatran / clopidogrel / dabigatran in randomized order
  Interventions: Drug: Clopidogrel; Drug: Dabigatran high dose; Drug: Dabigatran low dose
- Fixed sequence 2 (Experimental): intra-individual comparison with the fixed sequence of a single dose of 600mg clopidogrel alone and the combination of dabigatran 150 mg in steady state plus single dose of 600 mg clopidogrel
  Interventions: Drug: Clopidogrel; Drug: Dabigatran high dose

INTERVENTIONS:
Drug: Clopidogrel
Drug: Dabigatran high dose
Drug: Dabigatran low dose
  Arms: Crossover; Fixed sequence 1

SUMMARY:
The primary objective of the study (Main Part 2) was to investigate whether and to which extent a combination of multiple oral doses (steady state conditions) of 75 mg of clopidogrel q.d. (after a loading dose of 300 mg) and multiple doses of 150 mg of dabigatran etexilate b.i.d. at steady state affects pharmacokinetic and pharmacodynamic parameters of dabigatran etexilate and clopidogrel.

The objective of the preceding Pilot Part 1 of the study was to explore the effect of a single dose of 300 mg clopidogrel administered after multiple doses of 75 mg and 150 mg dabigatran had reached steady state, regarding safety as well as pharmacokinetic and pharmacodynamic parameters.

The Main Part 3 of the study moreover was to compare intra-individually the effects of a single dose of 600 mg clopidogrel with the same dose, 600 mg clopidogrel, given additionally to multiple doses of 150 mg dabigatran in steady state condition with respect to safety and pharmacokinetic and pharmacodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), body temperature, 12-lead electrocardiogram, clinical laboratory tests
2. Age ≥18 and Age ≤40 years
3. Body mass index (BMI) ≥18.5 and ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. Any gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Subjects who in the investigator's judgement are perceived as having an increased risk of bleeding, for example because of:

   * Hemorrhagic disorders or bleeding diathesis
   * Occult blood in faeces or haematuria
   * Trauma or surgery within the last month or as long as an excessive risk of bleeding persists after these events, or planned surgery during trial participation
   * History of arteriovenous malformation or aneurysm
   * History of gastroduodenal ulcer disease, gastrointestinal haemorrhage and haemorrhoids
   * History of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding
   * Use of drugs that may interfere with haemostasis during trial conduct (e.g.acetyl salicylic acid or other non-steroidal anti-inflammatory drugs)
3. Relevant surgery of gastrointestinal tract
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Intake of any medication within four weeks of first dosing
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within four weeks prior to administration or during the trial, especially inhibitors or inducers of P-gp, CYP3A4 CYP2C9 or CYP2C19
10. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, nonsteroidal anti-rheumatic drugs, cumarin etc. within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within one month prior to administration or during the trial
12. Alcohol abuse (more than 60 g/day on a regular basis)
13. Drug abuse
14. Within 5 days of study medication no intake of grapefruit, grapefruit juice, or products containing grapefruit juice, Seville oranges, garlic supplements, or St. John's Worth
15. Blood donation (more than 100 mL within four weeks prior to administration)
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Male subjects do not agree to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the study. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two months)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma over one dosing interval at steady state) | up to 19 days
  for total dabigatran, clopidogrel and the inactive metabolite SR26334
AUC0-24,1 (area under the concentration-time curve of the analyte in plasma over one dosing interval after the loading dose) | up to 19 days
  for clopidogrel and the inactive metabolite SR26334
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) | up to 19 days
  for total dabigatran, clopidogrel and the inactive metabolite SR26334
Cmax,1 (maximum measured concentration of the analyte in plasma after the loading dose) | up to 19 days
  for total dabigatran, clopidogrel and the inactive metabolite SR26334
AUECIPA,0-24 (area under the effect curve of inhibition of platelet aggregation after the first dose of clopidogrel) | up to 19 days
Emax,IPA,0-24 (maximum percentage change - compared to baseline - in adenosine diphosphate-induced platelet aggregation after the loading dose of clopidogrel) | baseline, up to 19 days

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma from the time point 0 to the last quantifiable analyte plasma concentration) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
λz (terminal rate constant in plasma) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
t1/2 (terminal half-life of the analyte in plasma) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 8 weeks
  Clopidogrel and SR 26334 after the loading dose
Cmax, ss | up to 8 weeks
  free dabigatran after multiple dosing
AUCτ,ss | up to 8 weeks
  free dabigatran after multiple dosing
AUC0-tz,ss (area under the concentration-time curve of the analyte in plasma from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
tz,ss (time of last measureable concentration of the analyte in plasma within the dosing interval τ at steady state) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
tmax,ss (time from last dosing to the maximum concentration of the analyte in plasma at steady state on day 4) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
CL/F,ss (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
tmin,ss (time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
PTF (peak trough fluctuation) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
Cavg (average concentration of the analyte in plasma at steady state over a uniform dosing interval) | up to 8 weeks
  Clopidogrel and SR 26334; dabigatran (free and total) after multiple dosing
AUECt1-t2 (area under the effect curve (baseline corrected by ratio)) | up to 8 weeks
  for activated partial thromboplastin time, thrombin time and ecarin clotting time
ERmax (maximum effect ratio) | up to 8 weeks
  for activated partial thromboplastin time, thrombin time and ecarin clotting time
tmax (time to maximum effect) | up to 8 weeks
  for activated partial thromboplastin time, thrombin time and ecarin clotting time
Occurence of Adverse Events | up to 13 weeks
Assessment of Tolerability by investigator | up to 13 weeks